CLINICAL TRIAL: NCT07219303
Title: Dose Escalated CT-Based Adaptive Stereotactic Body Radiation Therapy Among Patients With Intermediate- and Favorable High- Risk Prostate Cancer (DE-CART)
Brief Title: Adaptive Radiation Therapy for Men With Intermediate- or High-Risk Prostate Cancer
Acronym: DE-CART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT-237; 25-1023 (Other: FCCC IRB)
Record Dates: First submitted 2025-09-16; First posted 2025-10-21 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: Adaptive; SBRT; Stereotactic body radiation therapy; QOL; Simultaneous integrated boost; SIB; Adenocarcinoma; Prostate Cancer; Prostate Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase I Dose escalated adaptive stereotactic body radiation therapy (SBRT) with a SIB (Experimental)
  Interventions: Radiation: adaptive stereotactic body radiation therapy (SBRT) with a SIB

INTERVENTIONS:
Radiation: adaptive stereotactic body radiation therapy (SBRT) with a SIB — This is a phase 1 dose finding study investigating escalated doses of adaptive prostate SBRT for patients with intermediate and favorable high risk prostate cancer. There will be a Bayseian Optimal Interval Design (BOIN) defining the dose escalation parameters and the dose will escalate as per Section 5.0. Treatment is 5 fractions every other day and will be expected to be typically completed in 2-3 calendar weeks.

SUMMARY:
The goal of this clinical trial is to evaluate if adaptive stereotactic body radiation therapy (SBRT) is a safe and effective way to treat prostate cancer in adults. It will assess the safety profile of adaptive SBRT over time.

The main questions this trial aims to answer are:

* What is highest dose of adaptive SBRT without causing serious side effects?
* Can adaptive SBRT more precisely targeting the prostate while reducing radiation exposure to nearby organs?
* What side effects do participants experience during treatment, right after treatment, and over the five years post-treatment?
* Can adaptive SBRT reduce urination-related side effects and support quality of life during and after treatment?

Participants will:

* Receive adaptive SBRT treatment every other day, for a total of 5 treatment sessions (called fractions). The full course of treatment typically takes 2 to 3 weeks.
* Have a follow-up phone call about 6 weeks after treatment to check on side effects and overall wellbeing.
* Visit the clinic for check-ups and tests:

  * At 90 days (about 3 months) after treatment
  * Then every 3 months for the first year
  * Then every 6 months after that

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically confirmed intermediate- and favorable high risk (AJCC 8th ed stage IIA-IIC) adenocarcinoma of the prostate.
2. Age > 18 years.
3. ECOG performance status ≤ 2
4. Prostate volume (segmented) ≤ 100 cc determined by MRI and/or US within 24 mo of treatment for patients not on ADT and within 6 mo for patients on prior ADT. A simulation MRI is acceptable.
5. Subjects must have had a pre-treatment diagnostic multiparametric MRI prostate (mpMRI) showing a PI-RADS3, 4 or 5 lesion or a 68Ga- or 18F-PSMA (TLX591-CDx or piflufolastat F18) PET/CT within 12 mo of study registration.
6. Baseline International Prostate Symptom Score (IPSS) is ≤ 15. Baseline alpha blocker use is allowed.
7. Subjects must have full capacity to understand and be willing to sign the informed consent document.

Exclusion Criteria:

1. Subjects must not be experiencing toxicity CTCAE grade ≥ 3 GU or GI toxicity at baseline.
2. Subjects must not be receiving any other investigational agents.
3. Subjects must not have had prior pelvic radiation therapy.
4. Subjects must not have node-positive disease.
5. Subjects must not have extraprostatic extension determined by MRI prostate within 24 mo of treatment. For patients receiving ADT, the prostate MRI must have been obtained prior to the start of ADT.
6. Subjects must not have had prior ablative therapies for prostate cancer including cryosurgery, HIFU and nanoknife.
7. Subjects with prior TURP or laser enucleation are eligible. However, patients that have undergone prior simple prostatectomy are excluded.
8. Subjects that are receiving other antineoplastic agents including methotrexate are ineligible. Subjects that have received prior ADT are eligible if they have received < 6 mo total of ADT, if last administration of ADT was > 6 mo prior to registration and serum total testosterone levels have recovered to at least 100 ng/dL. Subjects with prior cancer diagnoses are eligible provided that treatment was completed and no evidence of disease status achieved at least 2 years prior to study registration.
9. Subjects must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
10. Any condition or significant co-morbidity that prevents safe delivery of SBRT per the discretion of the treating physician(s).
11. Subjects with active inflammatory bowel disease or active collagen vascular disorder.
12. Subjects that cannot undergo prostate fiducial placement.
13. Subjects that cannot undergo rectal spacer placement are excluded. Please, note that a rectal spacer incorporating iodine or similar CT contrast is preferred. However, patients that are able to only have a non-contrast rectal spacer due to iodine allergy or similar contraindication remain eligible.
14. Subjects that cannot undergo prostate MRI.
15. Subjects with bilateral prosthetic hips will be excluded. Subjects with unilateral prosthetic hips will be eligible only if the initial treatment plan meets all target and normal tissue constraints without protocol violation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2033-08-01 (Estimated); Study Completion 2033-11-01 (Estimated)

PRIMARY OUTCOMES:
Severe (CTCAE grade ≥ 3) treatment-related (possibly, probably or definitely) toxicity occurring within 90 days of treatment. | From initiation of treatment to 90 days after end of treatment, for a duration of ~100 days.

SECONDARY OUTCOMES:
Biochemically progression free survival | From end of treatment to biochemical, local, regional or distant progression, or initiation of additional prostate cancer therapy or death, or end of follow up for a total of up to 5 years.
  Time from the end of treatment administration to biochemical progression (using Pheonix definition), local, regional, or distant progression, initiation of additional prostate cancer therapy, or death. Patients who are alive and have not experienced any progression or initiated any additional prostate cancer therapy by the end of follow up are considered censored.
Local failure free survival | From end of treatment to local progression or death or end of follow up for a total of up to 5 years.
  Time from the end of treatment administration to local progression or death. Patients who are still alive and have not had local progression by the end of follow up are considered censored.
PSA response | From end of treatment to end of follow-up for a total of up to 5 years.
  The PSA response will be assessed by the post-treatment PSA nadir and time to nadir.
The proportion of patients who have a decrease greater than or equal to the acute minimum clinically important difference (MID) in EPIC-26 scores among the urinary, bowel and sexual function domains at 3 and 6 months post-treatment compared to baseline | From enrollment to 6 months post-treatment.
The proportion of patients who have a decrease greater than or equal to the minimum clinically important difference (MID) in EPIC-26 scores among the urinary, bowel and sexual function domains at 1 and 2 years post-treatment compared to baseline. | From enrollment to 2 years post-treatment for a duration of ~ 2.5 years.
Distant metastasis free survival | From end of treatment to distant metastasis or death or end of follow up, for a total of up to 5 years.
  Time from the end of treatment administration to distant metastasis or death. Patients who are still alive and metastasis-free at the end of follow up are considered censored.
The proportion of patients who had at least one optimal treatment planning criteria not met, the number of criteria not met per patient, and the number of criteria not met per organ site. | From radiation simulation to end of treatment for a duration of 2-3 months.
  These proportions will be assessed in the overall population and per dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Hallman, MD, PhD, Principal Investigator — FCCC
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States